CLINICAL TRIAL: NCT04345809
Title: Effect of Prophylactic Prosthesis Placement With Versus Without Omega-3 at the Umbilical Trocar Level on Surgical Site Infection and Herniation After Laparoscopic Cholecystectomy in Patients With Risk Factors.
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Marta Bellón, FISABIO, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: AGHO MYL PRELIMI
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Melanocyte-Stimulating Hormones; Docosahexaenoic Acids

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A. MESH WITH OMEGA-3: Group A - 6.4-cm diameter circular prosthesis C-QUR V-Patch with an omega-3 coating
  Interventions: Procedure: MESH WHIT OMEGA-3
- GROUP B. MESH WITHOUT OMEGA-3: Group B - 6.4-cm diameter circular prosthesis BARD Hernia Patch , without omega-3 in its composition
  Interventions: Procedure: MESH WITHOUT OMEGA-3

INTERVENTIONS:
Procedure: MESH WHIT OMEGA-3 — Mesh placement with Omega-3 at the umbilical trocar level after laparoscopic cholecystectomy in patients with risk factors for SSI and eventration.
  Groups: GROUP A. MESH WITH OMEGA-3
Procedure: MESH WITHOUT OMEGA-3 — Mesh placement without Omega-3 at the umbilical trocar level after laparoscopic cholecystectomy in patients with risk factors for SSI and eventration.
  Groups: GROUP B. MESH WITHOUT OMEGA-3

SUMMARY:
TITLE:

Effect of prophylactic prosthesis placement with versus without omega-3 at the umbilical trocar level on surgical site infection and herniation after laparoscopic cholecystectomy in patients with risk factors.

OBJECTIVE: To evaluate whether the placement of a synthetic prosthesis with omega-3 in its composition at the level of the umbilical trocar after laparoscopic cholecystectomy versus the placement of a synthetic umbilical prosthesis without omega-3 in its composition decreases the rate of surgical site infection (SSI) and trocar site hernia (TSH) in patients with risk factors for infection and herniation.

DETAILED DESCRIPTION:
METHODS: A prospective study was conducted with 2 consecutive series of patients operated on for cholelithiasis who also had some of the following risk factors that increase the occurrence of SSI or TSH: BMI > 30 kg/m2, diabetes mellitus, age > 65 years and chronic obstructive pulmonary disease. A circular prosthesis with an omega-3 coating was placed in patients in group A, and a prosthesis without omega-3 in its composition was placed in patients in group B. The main variables evaluated were the occurrence of SSI and TSH.

ELIGIBILITY:
Inclusion Criteria:

The included patients were between the ages of 18 and 90 years, underwent elective laparoscopic cholecystectomy for symptomatic cholelithiasis and had one of the following risk factors that increase the occurrence of SSI or TSIH:

* Obesity: with a body mass index (BMI) > 30 kg/m2.
* Diabetes Mellitus (insulin dependent or who take oral antidiabetic drugs),
* Age > 65 years and
* COPD treated with inhalers.

Exclusion Criteria:

* Nonfulfillment of the inclusion criteria.
* Conversion to laparotomy during the surgical procedure
* Non-acceptance of participation in the study by the patient
* Loss to follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were between the ages of 18 and 90 years, underwent elective laparoscopic cholecystectomy for symptomatic cholelithiasis and had one of the following risk factors that increase the occurrence of SSI or TSIH, included in general surgery consultations.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
SSI | 1 year
  Surgical Site Infection.
TSIH | 1 year
  Trocar site incisional hernia.

IPD SHARING:
Plan to Share IPD: Undecided
All individual patient data may be used by other researchers in terms of advancing research in this field.

REFERENCES:
- [Background] Tomioka K, Murakami M, Fujimori A, Watanabe M, Koizumi T, Goto S, Otsuka K, Aoki T. Risk Factors for Transumbilical Wound Complications in Laparoscopic Gastric and Colorectal Surgery. In Vivo. 2017 Sep-Oct;31(5):943-948. doi: 10.21873/invivo.11151. PMID 28882963
- [Background] Bowler PG, Jones SA, Walker M, Parsons D. Microbicidal properties of a silver-containing hydrofiber dressing against a variety of burn wound pathogens. J Burn Care Rehabil. 2004 Mar-Apr;25(2):192-6. doi: 10.1097/01.bcr.0000112331.72232.1b. PMID 15091147
- [Background] Sanders D, Lambie J, Bond P, Moate R, Steer JA. An in vitro study assessing the effect of mesh morphology and suture fixation on bacterial adherence. Hernia. 2013 Dec;17(6):779-89. doi: 10.1007/s10029-013-1124-5. Epub 2013 Jun 19. PMID 23780573
- [Background] Lai NM, Chaiyakunapruk N, Lai NA, O'Riordan E, Pau WS, Saint S. Catheter impregnation, coating or bonding for reducing central venous catheter-related infections in adults. Cochrane Database Syst Rev. 2016 Mar 16;3(3):CD007878. doi: 10.1002/14651858.CD007878.pub3. PMID 26982376
- [Background] Minar E, Schillinger M. Innovative technologies for SFA occlusions: drug coated balloons in SFA lesions. J Cardiovasc Surg (Torino). 2012 Aug;53(4):481-6. PMID 22854528
- [Background] Fernandez-Gutierrez M, Olivares E, Pascual G, Bellon JM, San Roman J. Low-density polypropylene meshes coated with resorbable and biocompatible hydrophilic polymers as controlled release agents of antibiotics. Acta Biomater. 2013 Apr;9(4):6006-18. doi: 10.1016/j.actbio.2012.12.012. Epub 2012 Dec 20. PMID 23261925
- [Background] Chopra I. The increasing use of silver-based products as antimicrobial agents: a useful development or a cause for concern? J Antimicrob Chemother. 2007 Apr;59(4):587-90. doi: 10.1093/jac/dkm006. Epub 2007 Feb 16. PMID 17307768
- [Background] Maicas VT, Rochina IJ. [Linoleic acid emulsion on the peri-lesion skin of venal ulcers. Action and cicatrizant effect. Corpus study]. Rev Enferm. 2008 Apr;31(4):26-32. Spanish. PMID 18564784
- [Background] Iannitti DA, Hope WW, Norton HJ, Lincourt AE, Millikan K, Fenoglio ME, Moskowitz M. Technique and outcomes of abdominal incisional hernia repair using a synthetic composite mesh: a report of 455 cases. J Am Coll Surg. 2008 Jan;206(1):83-8. doi: 10.1016/j.jamcollsurg.2007.07.030. Epub 2007 Oct 18. PMID 18155572
- [Background] Justinger C, Slotta JE, Ningel S, Graber S, Kollmar O, Schilling MK. Surgical-site infection after abdominal wall closure with triclosan-impregnated polydioxanone sutures: results of a randomized clinical pathway facilitated trial (NCT00998907). Surgery. 2013 Sep;154(3):589-95. doi: 10.1016/j.surg.2013.04.011. Epub 2013 Jul 13. PMID 23859304
- [Background] Sugerman HJ, Kellum JM Jr, Reines HD, DeMaria EJ, Newsome HH, Lowry JW. Greater risk of incisional hernia with morbidly obese than steroid-dependent patients and low recurrence with prefascial polypropylene mesh. Am J Surg. 1996 Jan;171(1):80-4. doi: 10.1016/S0002-9610(99)80078-6. PMID 8554156
- [Background] Sauerland S, Korenkov M, Kleinen T, Arndt M, Paul A. Obesity is a risk factor for recurrence after incisional hernia repair. Hernia. 2004 Feb;8(1):42-6. doi: 10.1007/s10029-003-0161-x. Epub 2003 Sep 6. PMID 13680307
- [Background] Anthony T, Bergen PC, Kim LT, Henderson M, Fahey T, Rege RV, Turnage RH. Factors affecting recurrence following incisional herniorrhaphy. World J Surg. 2000 Jan;24(1):95-100;discussion 101. doi: 10.1007/s002689910018. PMID 10594211
- [Background] Comajuncosas J, Vallverdu H, Orbeal R, Pares D. [Trocar site incisional hernia in laparoscopic surgery]. Cir Esp. 2011 Feb;89(2):72-6. doi: 10.1016/j.ciresp.2010.08.007. Epub 2011 Jan 20. Spanish. PMID 21255770
- [Background] Arroyo A, Garcia P, Perez F, Andreu J, Candela F, Calpena R. Randomized clinical trial comparing suture and mesh repair of umbilical hernia in adults. Br J Surg. 2001 Oct;88(10):1321-3. doi: 10.1046/j.0007-1323.2001.01893.x. PMID 11578284
- [Background] Wang XC, Zhang D, Yang ZX, Gan JX, Yin LN. Mesh reinforcement for the prevention of incisional hernia formation: a systematic review and meta-analysis of randomized controlled trials. J Surg Res. 2017 Mar;209:17-29. doi: 10.1016/j.jss.2016.09.055. Epub 2016 Oct 4. PMID 28032555
- [Background] Tang Y, Zhang MJ, Hellmann J, Kosuri M, Bhatnagar A, Spite M. Proresolution therapy for the treatment of delayed healing of diabetic wounds. Diabetes. 2013 Feb;62(2):618-27. doi: 10.2337/db12-0684. Epub 2012 Oct 5. PMID 23043160
- [Background] Pereira JA, Pera M, Grande L. [Incidence of incisional hernia after open and laparoscopic colorectal cancer resection]. Cir Esp. 2013 Jan;91(1):44-9. doi: 10.1016/j.ciresp.2012.05.004. Epub 2012 Jul 4. Spanish. PMID 22769029
- [Background] Armananzas L, Ruiz-Tovar J, Arroyo A, Garcia-Peche P, Armananzas E, Diez M, Galindo I, Calpena R. Prophylactic mesh vs suture in the closure of the umbilical trocar site after laparoscopic cholecystectomy in high-risk patients for incisional hernia. A randomized clinical trial. J Am Coll Surg. 2014 May;218(5):960-8. doi: 10.1016/j.jamcollsurg.2014.01.049. Epub 2014 Feb 18. PMID 24680572
- [Background] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Background] Chanda W, Joseph TP, Guo XF, Wang WD, Liu M, Vuai MS, Padhiar AA, Zhong MT. Effectiveness of omega-3 polyunsaturated fatty acids against microbial pathogens. J Zhejiang Univ Sci B. 2018 Apr.;19(4):253-262. doi: 10.1631/jzus.B1700063. PMID 29616501
- [Background] Woodrow T, Chant T, Chant H. Treatment of diabetic foot wounds with acellular fish skin graft rich in omega-3: a prospective evaluation. J Wound Care. 2019 Feb 2;28(2):76-80. doi: 10.12968/jowc.2019.28.2.76. PMID 30767649
- [Background] Alam K, Jeffery SLA. Acellular Fish Skin Grafts for Management of Split Thickness Donor Sites and Partial Thickness Burns: A Case Series. Mil Med. 2019 Mar 1;184(Suppl 1):16-20. doi: 10.1093/milmed/usy280. PMID 30901429
- [Background] Brathwaite S, Latchana N, Esemuede I, Harzman A, Husain S. Risk Factors for Surgical Site Infection in Open and Laparoscopic Hartmann Closure: A Multivariate Analysis. Surg Laparosc Endosc Percutan Tech. 2017 Feb;27(1):51-53. doi: 10.1097/SLE.0000000000000365. PMID 28145967
- [Background] Alfonso-Sanchez JL, Martinez IM, Martin-Moreno JM, Gonzalez RS, Botia F. Analyzing the risk factors influencing surgical site infections: the site of environmental factors. Can J Surg. 2017 Jun;60(3):155-161. doi: 10.1503/cjs.017916. PMID 28234221
- [Background] Cheadle WG. Risk factors for surgical site infection. Surg Infect (Larchmt). 2006;7 Suppl 1:S7-11. doi: 10.1089/sur.2006.7.s1-7. PMID 16834549
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487